CLINICAL TRIAL: NCT03680287
Title: Effects of Sleep Disruption on Drug Response
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB00160629; R01DA048206 (NIH)
Record Dates: First submitted 2018-08-27; First posted 2018-09-21 (Actual); Last update posted 2025-07-07 (Actual); Status verified 2025-07

CONDITIONS: Low Back Pain, Recurrent; Healthy
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Uninterrupted Sleep (Active Comparator): Participants will be permitted to sleep without interruption for 8 hours.
  Interventions: Drug: Within-Subject test of blinded study medication
- Sleep Disruption (Experimental): Participants will be repeatedly awakened throughout the night according to a standardized protocol.
  Interventions: Drug: Within-Subject test of blinded study medication

INTERVENTIONS:
Drug: Within-Subject test of blinded study medication — On the day after each sleep condition (Uninterrupted Sleep and Sleep Disruption), participants will undergo multiple injections of study medication or placebo. This is a double-blind within-subject Phase II trial. As such, study medications must remain blinded. Participants may receive a medication from one or more of the following categories: prescription stimulants, prescription benzodiazepines, prescription opioids, prescription cannabinoids, over-the-counter medications, or placebo (saline). This study uses a within-subject design, such that participants serve as participants' own control.

SUMMARY:
The central scientific premise of the proposed study is that sleep disruption (SD) will influence individuals' subjective response to blinded medication administration. The investigators further believe these responses will vary among patients who have chronic low back pain (CLBP) vs. healthy controls, and that sex will moderate effects.

The proposed study evaluates whether CLBP patients' subjective responses to study medication administration are altered by SD. The investigators focus on two outcome domains: abuse liability (i.e., drug liking and valuation) and response to pain testing.

The investigators propose a mixed between-within randomized crossover human-laboratory experiment that investigates placebo-controlled effects of study medication on 1) abuse liability metrics (Drug Liking and Monetary Valuation) and 2) response to laboratory-evoked standardized pain measures, after one night of uninterrupted sleep (US) and again after one night of SD. The investigators will recruit both CLBP patients(*) and healthy controls (N = 60).

(*) We originally aimed to accrue 60 subjects with CLBP. However, we have been granted approval by the National Institute on Drug Abuse (NIDA) to reduce expectations for the target N for the CLBP cohort. We are no longer expected to recruit N=60 CLBP participants; this is a COVID-19 modification, and we are not required to re-do a power analysis.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria:

* 18-60 years old
* Less than 2 servings/day of caffeinated beverages and willing to discontinue 3 days prior to admission.

CLBP-Specific Inclusion Criteria:

* Have a physician-confirmed diagnosis of CLBP
* Report chronic low back pain.

Exclusion Criteria:

General Exclusion Criteria:

* BMI >40
* Significant medical or psychiatric morbidity within 6 months or lifetime history of bipolar disorder, psychotic disorder, seizure disorder
* Lifetime history of opioid use disorder
* Clinically significant abnormal complete blood count or comprehensive metabolic profile
* Any contraindicated medical condition (status asthmaticus; chronic obstructive pulmonary disease; reduced respiratory function; hypotension; hypertension; impairment of hepatic, pulmonary or renal functions; myxedema or hyperthyroidism; adrenocortical insufficiency; gastrointestinal obstruction; gall bladder disease; acute alcoholism; history of convulsive disorders; history of head injury)
* Current use of stimulants, opioids, benzodiazepines or other Central Nervous System (CNS) depressant
* Positive toxicology screen for opioids, stimulants, or recreational drugs
* Pregnancy or lactation
* Significant preadmission psychological distress.

Healthy Control and CLBP-Specific Exclusion Criteria:

* Report current medical/psychiatry history
* Report acute painful injury (within 3 months)
* Have a diagnosed chronic pain disorder.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 109 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2025-04-29 (Actual); Study Completion 2025-04-29 (Actual)

PRIMARY OUTCOMES:
Drug Liking as assessed by the Visual Analog Scale | up to 420 minute post-medication administration
  Visual Analog Scale (0-100), where 0=None and 100 = Extremely , in response to the question, "Do you like the drug?"
Heat Pain Threshold | up to 420 minute post-medication administration
  A thermode will gradually increase in temperature until the participant indicates when it "first feels painful". The outcome will be the temperature (degrees Celsius) at which the participant indicates they first feel pain.
Suprathreshold Tonic Heat Pain | up to 420 minute post-medication administration
  A painful temperature above threshold will be held tonically for a period of time, after which pain ratings are obtained on a 0-100 numerical rating scale, where 0 = "No Pain" and 100 = "Worst Pain Imaginable."
Monetary Valuation of Drug as assessed by the Drug vs. Money Multiple Choice Questionnaire | up to 420 minute post-medication administration
  Participants are presented with an array of choices (in dollar value) which they will compare to the option of receiving study drug. They will decide for each choice whether they would take the money (at that value) or the drug they received in the session. The outcome will be the "crossover point", which is the mean of the last price that the participant selected "drug" and the first price at which the participant selected "money".

SECONDARY OUTCOMES:
Good Drug Effects as assessed by the Visual Analog Scale | up to 420 minute post-medication administration
  Visual Analog Scale (0-100), where 0=None and 100 = Extremely , in response to the question, "Does the drug have any good effects?"
Bad Drug Effects as assessed by the Visual Analog Scale | up to 420 minute post-medication administration
  Visual Analog Scale (0-100), where 0=None and 100 = Extremely , in response to the question, "Does the drug have any bad effects?"
Level of "Highness" as assessed by Visual Analog Scale | up to 420 minute post-medication administration
  Visual Analog Scale (0-100), where 0=None and 100 = Extremely , in response to the question, "How high are you?"
Feeling of Sickness as assessed by Visual Analog Scale | up to 420 minute post-medication administration
  Visual Analog Scale (0-100), where 0=None and 100 = Extremely , in response to the question, "Does this drug make you feel sick?"
Clinical Pain | up to 420 minute post-medication administration
  This will be rated on a 0-100 Numerical Rating Scale, where 0 = "No Pain" and 100 = "Worst Pain Imaginable."

CONTACTS AND LOCATIONS:
Overall Officials: Michael T. Smith, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No